CLINICAL TRIAL: NCT05295745
Title: Multidisciplinary Intervention and Cognitive Remediation Therapy for Adults With Obesity: Study Protocol for a Randomized Controlled Trial
Brief Title: Multidisciplinary Intervention With Cognitive Remediation Therapy for Obese Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Autonoma de Ciudad Juarez (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIEB-2019-2-53
Record Dates: First submitted 2021-10-27; First posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Obesity
Keywords: Adult; obese; Cognitive remediation therapy; multidisciplinary
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: This study has two arms, experimental and control group. The first one will receive the treatment and the control group that does not receive it until the intervention group completes the treatment. Both groups will be measured before and after completion, with three months follow-up
Who Masked: Participant
Masking Description: The participants will not be notified about the intervention group or the control group and will be randomly assigned. The procedures of this study will be available only to the researchers, therapists, and the bioethics committee of the Autonomous University of Ciudad Juárez
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive remediation therapy and multidisciplinary intervention (Experimental): The participants (obese adults) in the experimental group will receive treatment with cognitive remediation therapy, nutritional and physical activity instruction through 18 weekly sessions of intervention.
  Interventions: Behavioral: Cognitive remediation therapy and multidisciplinary intervention
- Control (No Intervention): The control group participants will not receive the treatment until the experimental group participants complete the intervention and carry out the measurements

INTERVENTIONS:
Behavioral: Cognitive remediation therapy and multidisciplinary intervention — The Randomized Controlled Trial will comprise of multidisciplinary intervention and remediation cognitive therapy which will be conducted with obese diagnosed adults of 19-60 years old. The enrolled patients will be randomized in a two-arm control trial with repeated measures and follow-up of three months. The experimental group participants will receive the intervention, while the control group remains on a waiting list.
  Nutritional and physical activity plus cognitive remediation therapy sessions to improve the thoughts style, problem-solving, planning and organization, the emotions and body image are included
  Arms: Cognitive remediation therapy and multidisciplinary intervention

SUMMARY:
This study aims to describe the research procedures and treatment of a multidisciplinary intervention with cognitive remediation therapy for adults with obesity in a Randomized Controlled Trial. The changes will be measured before and after the intervention and three months follow-up. To evaluate them, psychometric, psychological, physiological, and physical activity tests will be taken.

DETAILED DESCRIPTION:
A randomized controlled clinical trial will be carried out, implementing a multidisciplinary intervention with cognitive remediation therapy on obese adults from Ciudad Juárez, Chihuahua, México. The efficacy of this therapy has been proved in several countries except México.

A randomized controlled trial (RCT) will be executed with both an experimental group and a control group, with repeated measures taken before and after intervention and follow ups of three months. The study will be simple blind and randomization technique will be use to one assign to one of the two conditions. The experimental group will first receive the intervention and once finalized, it will be applied to the control group.

The investigator's hypothesis suggests that an intervention of cognitive remediation therapy implemented simultaneously with nutritional education and physical activity improvement in body composition such a body mass index (BMI), waist ratio, body fat, blood chemistry, skin conductance, eating behavior, craving, and body image. An improvement is also expected for the values in the applied psychophysiological tests, the cognitive performance, as well as the eating behavior and physical activities of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Ages 19-60
* BMI >30
* BFP >25 (women)
* BFP >32 (Men)
* High waist circumference >88 cm (women)
* High waist circumference >94 cm (men)
* Signed informed consent

Exclusion Criteria:

* If the participant is enrolled in a weight control or physical exercise program.
* If the participant is under any medical psychological treatment
* If the participant is presenting any eating disorder, a thyroid or neurological diseases
* Pregnant women
* Unfinished procedures
* Less than 20% of assistance during the intervention

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-08 (Estimated); Primary Completion 2022-11-08 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in body mass index at week 18 and 3 months follow up | Baseline and week 18 with 3 months follow up
  Body Mass Index which will be determined as a participant weight in kg by his eight in meters² (kg/mts²). Basis will be the values set by World Health Organization
Changes from baseline in waist circumference at week 18 and 3 months follow up | Baseline and week 18 with 3 months follow up
  Waist ratio will mesure and expressed in centimeters. The individual will be measured in a straight position, from the narrowest part of the trunk, free of clothing, a flexible metric tape will be used, the middle part between the costal flange and the iliac crest serving as a reference point.
Changes from baseline in body fat at week 18 and 3 months follow up | Baseline and week 18 with 3 months follow up
  Will be recorded and determined through the Seca mBCA 525 body analysis monitor, which includes electronic stadimeter, weighing platform with a 300 kg. capacity, tactile monitor, automatic detection electrode system and electronic system for data recording through the Seca analyticsm BCA 115 software.
Changes from baseline in blood chemistry at week 18 and 3 months follow up | Baseline and week 18 with 3 months follow up
  To determine the levels for glucose and lipids the CardioCkek PA capilar measurer will be used for it provides fast blood chemistry values and measurements. Basis will be the values set by the Diabetes Latin American Association for Latin American populations which establishes as normal for both glucose and lipids, values larger than or equal to 100 mg/dl establishes as normal for both glucose and lipids, values larger than or equal to 100 mg/dl.
Changes from baseline in eating behavior at week 18 and 3 months follow up | Baseline and week 18 with 3 months follow up
  The eating behavior it will established through the 24 hour dietary recall method, recording a normal day's food consumption throughout the day. A format will be used describing the ingredients, type and quantity of food and the hour and location of consumption. This procedure allows learning the quantity of calories consumed and type of macro-nutrients.
Changes from baseline in craving at week 18 and 3 months follow up | Baseline and week 18 with 3 months follow up
  The Food Craving Questionnaire-Trait will be used in its Spanish version to measure the intensity with which the desire for eating presents itself. This scale assesses nine subscales: (1) plans and intentions for eating, (2) positive reinforcement anticipation that might result from eating, (3) relief anticipation regarding negative feelings state that result from eating, (4) lack of control over food, (5) thoughts or concerns about food, (6) craving as a physiological state, (7) emotions that might be felt before or during the craving for food or while eating, (8) craving trigger signs for food, (9) sense of guilt because of craving or for giving in to it.
Changes from baseline in body image at week 18 and 3 months follow up | Baseline and week 18 with 3 months follow up
  A body form questionnaire will be used, which consists of a 34-item scale that explore the body image's self-perception and allows for the evaluation of both the body image dissatisfaction and the worry for it. This scale has a Cronbach's alpha of .98

SECONDARY OUTCOMES:
Mental flexibility-changes from baseline in the classification card subscale of the Neuropsychological Battery of Executive Functions and Frontal Lobes | 18 weeks with 3 months follow-up
  The classification card subtest assesses the ability to generate a classification hypothesis and ability of changes criteria (mental flexibility). The score is calculated recording the correct responses and three types of error; normal error, perseverations, deferred perseverations and maintenance errors.
Inhibitory control-changes from baseline in the Stroop effect subscale of the Neuropsychological Battery of Executive Functions and Frontal Lobes | 18 weeks with 3 months follow up
  The inhibitory control measurement will be performed using the Stroop effect subscale in his both forms A and B, which evaluates the capability of inhibitory control. In both parts two types of errors and execution time are logged. The types of errors can be made are Stroop and Non-Stroop error.
Working memory-changes from baseline in working memory index scale of the Wechsler Adult Intelligence Scale | 18 weeks with 3 months follow up
  The working memory index is a comprised of subtests that assess simultaneous and sequential processing, attention and concentration. Are included two core subtests: digit span, arithmetic and a supplemental subtest, letter-number sequencing, retention of digits, arithmetic and succession of numbers and letters that provide an evaluation of the work memory, measuring the capability to receive information, learn it in the short term and operate with it to achieve an objective.
Working memory-changes from baseline in self-directed signaling subscale of the Neuropsychological Battery of Executive Functions and Frontal Lobes | 18 weeks with 3 months follow up
  The subscale to be used will be the one denominated as self-directed signaling which evaluates the capability to use the viso-spatial work memory to point in a self-directed manner a set of figures and no repeat or omit any. The maximum score to achieve in this test is 25.
Working memory-changes from baseline in ordering of words subscale of the the Neuropsychological Battery of Executive Functions and Frontal Lobes | 18 weeks with 3 months follow up
  The subscale for alphabetical ordering of words will be used, which calculates the capability to manipulate and mentally order the verbal information contained in the working memory. The score is calculated based on the following aspects: Rehearsal number in which the list is played correctly, perseverance of words that the person repeats more than once, intrusions; words that mention but are not on the list, orders errors, words whose initial vowel or consonant does not correspond, and if the subject does not remember any words in the first trial.
Processing speed-changes from baseline in processing speed index scale of the Wechsler Adult Intelligence Scale | 18 weeks with 3 months follow up
  The processing speed index that will be used includes subtest measure the speed and graphomotor processing, includes two core subtests: symbol search and coding, and one supplemental subtest cancellation. Measurement of the processing speed is performed through the fast and correct response ability of those tasks that require observation and discrimination. For this purpose, the subscales denominated as symbols search, codes and cancellation will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Loya Yolanda, PhD, Principal Investigator — Universidad Autónoma de CIudad Juárez

IPD SHARING:
Plan to Share IPD: Yes
Will be published in index journals
Supporting Information: Study Protocol
Time Frame: December 2022
Access Criteria: Cognitive Remediation Therapy adult obesity

REFERENCES:
- [Background] Smith E, Hay P, Campbell L, Trollor JN. A review of the association between obesity and cognitive function across the lifespan: implications for novel approaches to prevention and treatment. Obes Rev. 2011 Sep;12(9):740-55. doi: 10.1111/j.1467-789X.2011.00920.x. No abstract available. PMID 21991597
- [Background] ALAD (2019). Latin American Diabetes Association. ALAD Guidelines concerning the Diagnosis, Control and Treatment of Type 2 Mellitus Diabetes with Medicine based on Evidence 2019 Edition. Latin American Diabetes Association Magazine ISSN: 2248-6518 México: Permanyer https://www.revistaalad.com/guias/5600AX191_guias_alad_2019.pdf
- [Background] Allom V, Mullan B, Smith E, Hay P, Raman J. Breaking bad habits by improving executive function in individuals with obesity. BMC Public Health. 2018 Apr 16;18(1):505. doi: 10.1186/s12889-018-5392-y. PMID 29661241
- [Background] Batterink L, Yokum S, Stice E. Body mass correlates inversely with inhibitory control in response to food among adolescent girls: an fMRI study. Neuroimage. 2010 Oct 1;52(4):1696-703. doi: 10.1016/j.neuroimage.2010.05.059. Epub 2010 May 25. PMID 20510377
- [Background] Cabas Hoyos, K., González Bracamonte Y. and Mendoza Álvarez C. (2017). Executive Functioning and Depression in college students with normoweight, overweight and obesity Type 1. Psychological Reports 18 (1) 133-144 https://doi.org/10.18566/infpsic.v18n1a07
- [Background] Camacho Laraña, M., Alcalá Pérez, V. and Alcalá S.N. (2020). Gender differences in patients with morbid obesity tributary to bariatric surgery. Psychopathology and Clinical Psychology Magazine. ISSN: 1136-5420 doi:10.5944/rppc.vol.20.number.3.2015.15892 Spain: Spanish Association of Clinical Psychology and Psychopathology
- [Background] Carretero Gomez J, Ena J, Arevalo Lorido JC, Segui Ripoll JM, Carrasco-Sanchez FJ, Gomez-Huelgas R, Perez Soto MI, Delgado Lista J, Perez Martinez P; en representacion del grupo de trabajo de Diabetes, Obesidad y Nutricion de la Sociedad Espanola de Medicina Interna. Obesity is a chronic disease. Positioning statement of the Diabetes, Obesity and Nutrition Workgroup of the Spanish Society of Internal Medicine (SEMI) for an approach centred on individuals with obesity. Rev Clin Esp. 2020 Jul 25:S0014-2565(20)30180-6. doi: 10.1016/j.rce.2020.06.008. Online ahead of print. English, Spanish. PMID 32723530
- [Background] Chao A, Grilo CM, White MA, Sinha R. Food cravings, food intake, and weight status in a community-based sample. Eat Behav. 2014 Aug;15(3):478-82. doi: 10.1016/j.eatbeh.2014.06.003. Epub 2014 Jun 18. PMID 25064302
- [Background] Dohle S, Diel K, Hofmann W. Executive functions and the self-regulation of eating behavior: A review. Appetite. 2018 May 1;124:4-9. doi: 10.1016/j.appet.2017.05.041. Epub 2017 May 25. PMID 28551113
- [Background] Flores Lázaro, J.C., OstroskyShejet, F. and Gutiérrez Loxano, A. (2014). Neuropsychological Development of frontal lobes and executive functions. Editorial/Publisher: The Modern Manual México
- [Background] Gómez Puente, J.M. y Martínez Marcos, M. (2017). Overweight and Obesity: Efficiency of interventions in adults. Clinical Nursing 28(1) 65-74 ISSN: 1130-8621 Spain: Elsevier https: doi.org/10.1016/j.enfcli.201 7.06.005
- [Background] González, M. (2018). Role of executive functions in comprehending food intake. Answers or voids? Gastroenterology Venezuelan Society Magazine Vol.72 Númber 2 pages 38-43 ISSN: 2477-975X On line: https://www.researchgate.net/publication/334045971_Rol_de_las_funcion
- [Background] Guarch Domènech, J. y Navarro Odriozola, V. (2016) Cognitive Psychotherapies. Biological Psychiatry. 23 (S1): 40-45 ISSN: 1134-5934 Spain: Elsevier and Spanish Society of Biological Psychiatry.
- [Background] Hernández Sampieri, R., Fernández Collado, C., y Baptista Lucio, P. (2014). Methodology of Research. México: Trillas Publisher/Editorial
- [Background] INSP National Institute of Public Health. Results Report of the National Health and Nutrition Survey (ENSANUT) 2018. México: National Institute of Public Health. On Line: https://ensanut.insp.mx/encuestas/ensanut2018/informes.php
- [Background] Lafuente, M.D. (2012). Cognitive Behavioral Treatment of Obesity Eating Behavior Disorders (14) 1490-1504 ISSN: 1699-7611 Spain: Behavioral Sciences Institute On Line: https://dialnet.unirioja.es/servlet/articulo?codigo=6250628
- [Background] Marin-Soto MD, Leon CV, Perez-Vielma NM, Castillo-Ramirez M, Miliar-Garcia A, Murillo-Tovar MM, Mendez-Pena B, Aguilera-Sosa VR. Intense craving for appetizing foods: validation and standardization of the Food Cravings Questionnaire-Trait in Mexico. Gac Med Mex. 2020;156(1):27-33. doi: 10.24875/GMM.19005358. PMID 32026878
- [Background] Meza Peña, C. y Pompa-Guajardo, E.G. (2016). Gender, obesity and self-concept in a teen sample in México. Sports Sciences International Magazine 44 (12) 137-148. ISSN:1885-3137 Spain: Editorial/Publisher Ramón Cantó Alcaraz On Line: http://www.redalyc.org/articulo.oa?id=71044746005
- [Background] Navarro Santos, F. (2014) Body Image Construction for Overweight Women. Guillén Riebeling, The Modern Manual, A.S. of V.C.
- [Background] Polo García, D. (2014). Relationship between food anxiety constructos, impulsiveness and sensibility towards the rewards in a college population (master's thesis) Jaén College, Andalucía, Spain.
- [Background] Raman J, Hay P, Smith E. Manualised Cognitive Remediation Therapy for adult obesity: study protocol for a randomised controlled trial. Trials. 2014 Nov 4;15:426. doi: 10.1186/1745-6215-15-426. PMID 25370364
- [Background] Raman J, Hay P, Tchanturia K, Smith E. A randomised controlled trial of manualized cognitive remediation therapy in adult obesity. Appetite. 2018 Apr 1;123:269-279. doi: 10.1016/j.appet.2017.12.023. Epub 2017 Dec 24. PMID 29278718
- [Background] Ramírez Molina, M.J. (2017). Body Image, body satisfaction, specific auto-efficiencies and risk and health behaviors to improve body image (doctoral thesis). University of Granada, Granada Spain. https://hera.ugr.es/tesisugr/26765640.pdf
- [Background] Ríos Saldaña, M.R. Rodríguez Soriano, N.Y. and Álvarez Gasca, M.A. (2014). Incidence of Obesity, risks factors and emotional problems in college students. Psychology of Obesity Life Spheres Multidiscipline and complexity 63-74 México: The Modern Manual, A.S of V.C.
- [Background] Risco, L. y Aros, C. (2019). Mood, nutrition and craving disorders. Chilean Journal of neuropsychiatry. 57 (30) 295-305 ISSN: 0717:9227 Chile: Neurology, Psychiatry and Neurology Society.
- [Background] Salvador Castell, G., Serra Majem, L. and Ribas Barba, L. (2015). What and how much do we eat? The 24 hour remember method. Spanish Magazine for Community Nutrition 21 (Suppl. 1): 42-44 ISSN: 1135-3074 Spain: Spanish Society for Community Nutrition and Latin american Group for Community Nutrition. Doi10.14642/RENC.2015.21.sup1.5049
- [Background] Segura, M., Roncero, M., Oltra Cucarella, J., Blasco, L., Ciscar, S., Portillo, M., Malea, A., Espert, R. y Perpiñá, C. (2017). Cognitive remediation Training and emotional abilities in a group format for patients with obesity: A pilot study. Psychopathology and Clinical Psychology Magazine. Vol.22 127-138 doi: 10.5944/rppc
- [Background] Shama Levy, T., Villalpando-Hernández, S. y Rivera-Dommarco, J. (2006). Procedure's Manual for nutrition projects. Public Health National Institute. On line: http://www.salud.gob.mx/unidades/cdi/documentos/proy_nutricion.pdf
- [Background] Smith, E., Hay, P. y Raman, J. (2014). Cognitive Remediation Therapy for obesity. En Tchanturia, K. Cognitive Remediation Therapy (CRT) for Eating and Weigth Disorders 176-190 England: Routledge
- [Background] Sociedad Mexicana de Psicología, Código ético del psicólogo. [Mexican Society of Psychology (2010). Ethical Code for the Psychologist México], Trillas, Ciudad de México, México
- [Background] Tchanturia, K., Davies, H., Reeder, C. y Wykes, T., (2012). Cognitive Remediation Therapy for Anorexia Nervosa. Translation by López, C., Escobar, T. and Carral, L.
- [Background] Genders R, Tchanturia K. Cognitive remediation therapy (CRT) for anorexia in group format: a pilot study. Eat Weight Disord. 2010 Dec;15(4):e234-9. doi: 10.1007/BF03325304. PMID 21406946
- [Background] Torres V, Castro Sanchez AM, Mataran Penarocha GA, Lara Palomo I, Aguilar Ferrandiz ME, Moreno Lorenzo C. [Benefits of cognitive behavior therapy and acupressure therapy in obese patients: a randomized clinical trial]. Nutr Hosp. 2011 Sep-Oct;26(5):1018-24. doi: 10.1590/S0212-16112011000500015. Spanish. PMID 22072347
- [Background] Vázquez Arévalo, R., Galán Julio, J., López Aguilar, X., Alvarez Rayón, G.L., Marcilla Díaz, J.M., Caballero Romo, A. and Unikel Santoncini C. (2011). Validity of Body Shape Questionnaire (BSQ) in Mexican Women. Mexican Magazine for Eating Disorders Vol. 2 pages. 45-52 ISSN: 2007-1523 México: Autonomous National University of México
- [Background] Verdejo-Garcia A, Bechara A. [Neuropsychology of executive functions]. Psicothema. 2010 May;22(2):227-35. Spanish. PMID 20423626
- [Background] Weschler, D. (2013). WAIS-IV Weschler's Intelligence Scale ISBN: 91-100 México: The Modern Manual.
- [Background] WHO World Health Organization. 10 facts about obesity. On Line: https://www.who.int/features/factfiles/obesity/es/, https://www.who.int/es/news- room/fact-sheets/detail/obesity-and-overweight
- [Background] WHO World Health Organization. GPAQ Analysis Guide On Line: https://www.who.int/ncds/surveillance/steps/resources/GPAQ_Analysis_Guide.pdf